CLINICAL TRIAL: NCT05769751
Title: A Multicenter, Non-interventional Retrospective Study to Describe the Real-world Treatment Patterns and Associated Outcomes in Patients of China With HER2-positive Unresectable or Metastatic Breast Cancer
Brief Title: A Study to Describe the Real-world Treatment Patterns and Associated Outcomes in Patients of China With HER2-positive Unresectable or Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DSCN-EHT-NIS-BC001
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: HER2-positive Breast Cancer
Keywords: HER2-positive Breast Cancer; Real-world study; Treatment patterns
MeSH Terms: interventions — Electronic Health Records; Hospital Information Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Electronic medical record and hospital information system or other available resources — This is a non-interventional study. No study medication will be provided to the participants.

SUMMARY:
This is a multicenter, non-interventional, retrospective, real-world study that enrolled patients diagnosed with HER2-positive unresectable or metastatic breast cancer. This study will be conducted to understand the treatment pattern and sequencing of therapies, survival outcomes, and associated burden of toxicities with line of treatment in the real world.

DETAILED DESCRIPTION:
The treatment landscape has changed dramatically with the lack of real-world evidence for usage and the efficacy of newly approved drugs in China. This multicenter, retrospective, non-interventional study will include patients newly diagnosed with HER2-positive unresectable or metastatic breast cancer, or first recurrent from early breast cancer.

The primary objective of this real-world study is to describe the treatment patterns of HER2-positive unresectable or metastatic breast cancer in China. Secondary objectives will include describing the demographic and clinicopathological characteristics of patients, efficacy of different treatment regimens, treatment options and efficacy of brain metastases, and safety and tolerability of different treatment regimens in patients with HER2-positive unresectable or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age at the time of diagnosis of unresectable or metastatic breast cancer
* Participants with first diagnosis of unresectable or metastatic breast cancer, or first recurrence of HER2-positive breast cancer since January 1, 2020. Participants were eligible if they were HER2-positive in the early operable stage and HER2-negative in the advanced stage. HER2 positive was defined with the reference to the Chinese guidelines for HER2 positive breast cancer at the time of testing
* Participants have received at least one systemic therapy for advanced breast cancer

Exclusion Criteria:

* Participants with concomitant cancer at the time of diagnosis of HER2-positive unresectable or metastatic breast cancer, except for the non-metastatic non-melanoma skin cancers, or in situ or benign neoplasms; a cancer is considered concomitant if it occurs within 5 years of HER2-positive breast cancer diagnosis.
* Participants who are/were currently/previously enrolled in a clinical trial and have not been unblinded during the data collection interval of the study
* Participants with critical missing data from their medical records or other patients deemed by the investigator to be ineligible for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be participants with a first diagnosis of HER2-positive unresectable or metastatic breast cancer or first recurrence between January 1, 2020 and August 31, 2022, who have at least one record of late systemic therapy, and were followed up until August 31, 2022. The study will be implemented at 4-6 top hospitals in Tier 1/2 cities spanning across China.
  Patient data will be retrospectively collected using the electronic medical record and hospital information system or other available resources, including laboratory test results, imaging, pathology reports, medical records, surgical records, prescription diagnoses, inpatient visits and hospitalizations.
Sampling Method: Non-Probability Sample
Enrollment: 865 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Receiving Each Regimen in Each Treatment Line | Assessed over a 2 year, 8 month time period
Treatment Sequence Since the Time of Diagnosis of HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
Percentage of Participants Receiving Endocrine Therapy if Breast Cancer is Hormone Receptor Positive | Assessed over a 2 year, 8 month time period
Percentage of Participants Receiving Local and Regional Treatment for Metastasis (Radiotherapy and/or Surgery) and Osteoprotective Therapy | Assessed over a 2 year, 8 month time period

SECONDARY OUTCOMES:
Percentage of Participants With HER2-positive Unresectable or Metastatic Breast Cancer, Based on Demographic and Clinicopathological Characteristics | Assessed over a 2 year, 8 month time period
Real-world Progression-free Survival (rwPFS) in Participants With HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
  Real-world progression-free survival (rwPFS) is defined as the time from initiation of treatment to disease progression or death due to any cause.
Time to Next Treatment (TTNT) in Participants With HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
  Time to next treatment is defined as the time from initiation of a systemic therapy to the date of initiation of the first subsequent systemic therapy regimen or death.
Duration of Treatment (DoT) in Participants With HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
  Duration of treatment is defined as the length of time a patient is treated.
Real-world Objective Response Rate (rwORR) in Participants With HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
  Real-world objective response rate is defined as the percentage of participants who have a partial response or complete response to treatment within a certain period of time.
Real-world Disease Control Rate (rwDCR) in Participants With HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
  Real-world disease control rate is defined as the percentage of participants with advanced or metastatic cancer who have achieved complete response, partial response, and stable disease.
Real-world Duration of Response (rwDoR) in Participants With HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
  Real-world duration of response is defined as the time from randomization to disease progression or death in participants who achieve complete or partial response.
Percentage of Participants With Brain Metastases Per Line of Treatment in Participants With HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
Percentage of Participants With HER2-positive Unresectable or Metastatic Breast Cancer, Based on Clinical Characteristics of Brain Lesions | Assessed over a 2 year, 8 month time period
Percentage of Participants Receiving Radiotherapy or Surgery in Participants With HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
Treatment Pattern After Diagnosis of Brain Metastases in Participants With HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
Real-world Progression-free Survival (rwPFS) After Diagnosis of Brain Metastases in Participants With HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
  Real-world progression-free survival (rwPFS) is defined as the time from initiation of treatment to disease progression or death due to any cause.
Time to Next Treatment (TTNT) After Diagnosis of Brain Metastases in Participants With HER2-positive Unresectable or Metastatic Breast Cancer | Assessed over a 2 year, 8 month time period
  Time to next treatment is defined as the time from initiation of a systemic therapy to the date of initiation of the first subsequent systemic therapy regimen or death.
Percentage of Participants With Adverse Events (AE) Leading to Treatment Discontinuation or Dose Modification | Assessed over a 2 year, 8 month time period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Daiichi Sankyo
Locations (5):
- China (5):
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan
  - Liaoning Cancer Hospital, Shenyang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No